CLINICAL TRIAL: NCT00203749
Title: NIMH Project Accept: A Phase III Randomized Controlled Trial of Community Mobilization, Mobile Testing, Same-Day Results, and Post-Test Support for HIV in Sub-Saharan Africa and Thailand
Brief Title: Community Mobilization, Mobile Testing, Same-Day Results, and Post-Test Support for HIV in Sub-Saharan Africa and Thailand
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); HIV Prevention Trials Network (Network)
Responsible Party: Principal Investigator, Thomas J. Coates, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U01MH066701 (NIH); U01MH066701 (NIH); U01MH066687 (NIH); U01MH066688 (NIH); U01MH066702 (NIH); DAHBR 9A-ASPG
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: HIV; Testing; Counseling
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention communities will receive the community-based VCT intervention community mobilization, mobile VCT, and post-test support services), as well as standard clinic-based VCT
  Interventions: Behavioral: Community-Based HIV VCT
- 2 (Active Comparator): Comparison communities will receive standard clinic-based VCT
  Interventions: Behavioral: Standard clinic-based VCT

INTERVENTIONS:
Behavioral: Community-Based HIV VCT — COMMUNITY MOBILIZATION. This component of the intervention uses community outreach to enhance the uptake of VCT, thus increasing the rate of HIV testing and frequency of discussions about HIV and reducing stigma through community education and mobilization.
  EASY ACCESS TO VCT. This component is designed to remove practical barriers and increase safety of VCT. Mobile vans or temporary units set up at local community sites will provide free, anonymous VCT in specific, chosen sites where people gather, such as market areas, shopping centers, and community centers.
  POST-TEST SUPPORT SERVICES. This component is designed to build psychosocial support to improve the quality of life for individuals diagnosed with HIV. The expected outcomes include a reduction in social harm, an increase in social support through disclosure to those most likely to provide support, and a reduction in internalized stigma. Social support should also decrease the behavioral risk of further transmission.
  Arms: 1
Behavioral: Standard clinic-based VCT — Control communities will receive Standard Clinic-Based VCT (SVCT) instead of the community-based VCT (CBVCT) intervention. Each of these communities will have access to SVCT that reflects local access to health care. The training for VCT counselors will be the same in the CBVCT and SVCT communities; however, no active recruitment for participation in the SVCT services will be made beyond the standard procedures of each clinic for informing patients of services (e.g., telling individual patients that VCT is available, posting of a flyer in the clinic announcing VCT availability, etc). As such, no active outreach or community mobilization will be conducted by the study staff in the SVCT settings (although it is possible that such activities will occur due to local initiative).
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a combination of clinic- and community-based voluntary counseling and testing programs in preventing HIV in African and Thai communities.

DETAILED DESCRIPTION:
NIMH Project Accept is an HIV prevention trial in which 48 communities (10 in Tanzania [Kisarawe], 8 in Zimbabwe [Mutoko], 8 in South Africa/Vulindlela, 8 in South Africa/Soweto and 14 in Thailand [Chiang Mai]) are being randomized to receive either a community-based HIV voluntary counseling and testing (CBVCT) intervention plus standard clinic-based VCT (SVCT), or SVCT alone. The CBVCT intervention has three major strategies: (1) to make VCT more available in community settings; (2) to engage the community through outreach; and (3) to provide post-test support. These strategies are designed to change community norms and reduce risk for HIV infection among all community members, irrespective of whether they participated directly in the intervention.

A community-level intervention based on modifying community norms can change the environmental context in which people make decisions about HIV risk, and has the potential to alter the course of the HIV epidemic in developing countries. This is the first international randomized controlled Phase III trial to determine the efficacy of a behavioral/social science intervention with an HIV incidence endpoint.

ELIGIBILITY:
Inclusion Criteria:

Baseline Assessment:

Persons may be included in the baseline behavioral assessment if they meet all of the following criteria:

* Reside in a community selected for the study
* Are randomly selected and invited to participate from households that are themselves randomly selected and invited to participate
* Aged 18-32 years
* Has lived in the community at least 4 months in the past year
* Sleeps regularly in their household at least 2 nights per week
* Able and willing to provide verbal informed consent

Qualitative Cohort:

Persons may be included in the qualitative cohort if they meet all of the following criteria:

* Participated in the baseline behavioral assessment
* Aged 18-32 years at enrollment
* Have not been away from the community for more than two months at a time in the last two years
* Able and willing to provide written informed consent

Intervention:

Persons may access community-based counseling and testing (in CBVCT communities) through the study if they meet all of the following criteria:

* >16 years of age
* Able and willing to provide verbal informed consent

Persons may access post-test support through the study if they meet all of the following criteria:

* >16 years of age
* Able and willing to provide verbal informed consent
* Proof of having been tested for HIV at a Project Accept CBVCT venue, irrespective of test result

Control:

Persons may access standard clinic-based counseling and testing (in both SVCT and CBVCT communities) through the study if they meet all of the following criteria:

* >16 years of age
* Able and willing to provide verbal informed consent

Post-Intervention Assessment:

Persons may be included in the post-intervention assessment if they meet all of the following criteria:

* Reside in a community selected for the study
* Are randomly selected to be offered to participate from households that are themselves randomly selected to be offered to participate
* Aged 18-32 years
* Has lived in the community at least 4 months in the past year
* Sleeps regularly in their household at least 2 nights per week
* Able and willing to provide informed consent (written for biological assessment; verbal for behavioral assessment)

Exclusion Criteria:

Baseline Assessment:

Persons will be excluded from the baseline behavioral assessment if they meet any of the following criteria:

* Are not a member of the study community or are not randomly selected to be offered to participate
* Are below 18 or above 32 years of age
* Has not lived in the community at least 4 months in the past year
* Does not sleep regularly in their household at least 2 nights per week
* Have an obvious psychological/psychiatric disorder that would invalidate the informed consent process or otherwise contraindicate participation in the assessment

Qualitative Cohort:

Persons will be excluded from the qualitative cohort if they meet any of the following criteria:

* Not a participant in the baseline behavioral assessment
* Less than 18 or greater than 32 years of age at enrollment
* Have been away from the community for more than two months at a time in the last two years
* Demonstrate signs of being visibly distraught, emotionally unstable, or under the influence of psychoactive agents that would invalidate the consent process or otherwise contraindicate participation in the qualitative assessment
* Have concrete plans to leave the community, thus removing possibility of follow up

Intervention:

Persons will be excluded from accessing counseling and testing (CBVCT) through the study (and will be referred to existing alternate services) if they meet any of the following criteria:

* <16 years of age
* Have an obvious psychological/psychiatric disorder that would invalidate the informed consent process or otherwise contraindicate participation

Persons will be excluded from accessing post-test support through the study (and will be referred to existing alternate services) if they meet any of the following criteria:

* <16 years of age
* Have an obvious psychological/psychiatric disorder that would invalidate the informed consent process or otherwise contraindicate participation

Control:

* <16 years of age
* Have an obvious psychological/psychiatric disorder that would invalidate the informed consent process or otherwise contraindicate participation

Post-Intervention Assessment:

Persons will be excluded from the post-intervention assessment if they meet any of the following criteria:

* Are not a member of the study community or are not randomly selected to be offered to participate
* Are below 18 or above 32 years of age
* Has not lived in the community at least 4 months in the past year
* Does not sleep regularly in their household at least 2 nights per week
* Have an obvious psychological/psychiatric disorder that would invalidate the informed consent process or otherwise contraindicate participation in the assessment

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 192814 (Actual)
Dates: Start 2004-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of recent HIV infection | Measured at Year 3

SECONDARY OUTCOMES:
Less HIV risk behavior | Measured at Year 3
Higher rates of HIV testing | Measured at Year 3
More favorable social norms regarding HIV testing | Measured at Year 3
More frequent discussions about HIV | Measured at Year 3
More frequent disclosure of HIV status | Measured at Year 3
Less HIV-related stigma | Measured at Year 3
Fewer HIV-related life events | Measured at Year 3

CONTACTS AND LOCATIONS:
Overall Officials: David Celentano, ScD, MHS, Principal Investigator — Johns Hopkins University; Thomas J Coates, PhD, Principal Investigator — University of California, Los Angeles; Stephen F Morin, PhD, Principal Investigator — University of California, San Francisco; Michael Sweat, PhD, Principal Investigator — Medical University of South Carolina; Michal Kulich, PhD, Principal Investigator — Charles University, Czech Republic; Deborah Donnell, PhD, Principal Investigator — SCHARP, Fred Hutchinson Cancer Research Center; Linda Richter, PhD, Principal Investigator — Human Sciences Research Council; Glenda Gray, MBBCH, FCPaeds(SA), Principal Investigator — University of Witwatersrand, South Africa; Jessie Mbwambo, MD, Principal Investigator — Muhimbili University; Alfred Chingono, MSc, Principal Investigator — University of Zimbabwe; Suwat Chariyalertsak, MD, DrPH, Principal Investigator — Chiang Mai University
Locations (5):
- South Africa (2):
  - University of the Witwatersrand, Soweto, Johannesburg, Gauteng
  - Human Sciences Research Council, Pietermaritzburg, KwaZulu-Natal
- Muhimbili University, Dar es Salaam, Tanzania
- Chiang Mai University, Chiang Mai, Chiang Mai, Thailand
- University of Zimbabwe, Harare, Zimbabwe

REFERENCES:
- [Derived] Coates TJ, Kulich M, Celentano DD, Zelaya CE, Chariyalertsak S, Chingono A, Gray G, Mbwambo JK, Morin SF, Richter L, Sweat M, van Rooyen H, McGrath N, Fiamma A, Laeyendecker O, Piwowar-Manning E, Szekeres G, Donnell D, Eshleman SH; NIMH Project Accept (HPTN 043) study team. Effect of community-based voluntary counselling and testing on HIV incidence and social and behavioural outcomes (NIMH Project Accept; HPTN 043): a cluster-randomised trial. Lancet Glob Health. 2014 May;2(5):e267-77. doi: 10.1016/S2214-109X(14)70032-4. Epub 2014 Apr 8. PMID 25103167
- [Derived] Laeyendecker O, Piwowar-Manning E, Fiamma A, Kulich M, Donnell D, Bassuk D, Mullis CE, Chin C, Swanson P, Hackett J Jr, Clarke W, Marzinke M, Szekeres G, Gray G, Richter L, Alexandre MW, Chariyalertsak S, Chingono A, Celentano DD, Morin SF, Sweat M, Coates T, Eshleman SH. Estimation of HIV incidence in a large, community-based, randomized clinical trial: NIMH project accept (HIV Prevention Trials Network 043). PLoS One. 2013 Jul 11;8(7):e68349. doi: 10.1371/journal.pone.0068349. Print 2013. PMID 23874597
- [Derived] Piwowar-Manning E, Fiamma A, Laeyendecker O, Kulich M, Donnell D, Szekeres G, Robins-Morris L, Mullis CE, Vallari A, Hackett J Jr, Mastro TD, Gray G, Richter L, Alexandre MW, Chariyalertsak S, Chingono A, Sweat M, Coates T, Eshleman SH. HIV surveillance in a large, community-based study: results from the pilot study of Project Accept (HIV Prevention Trials Network 043). BMC Infect Dis. 2011 Sep 24;11:251. doi: 10.1186/1471-2334-11-251. PMID 21943026
- [Derived] Sweat M, Morin S, Celentano D, Mulawa M, Singh B, Mbwambo J, Kawichai S, Chingono A, Khumalo-Sakutukwa G, Gray G, Richter L, Kulich M, Sadowski A, Coates T; Project Accept study team. Community-based intervention to increase HIV testing and case detection in people aged 16-32 years in Tanzania, Zimbabwe, and Thailand (NIMH Project Accept, HPTN 043): a randomised study. Lancet Infect Dis. 2011 Jul;11(7):525-32. doi: 10.1016/S1473-3099(11)70060-3. Epub 2011 May 3. PMID 21546309